CLINICAL TRIAL: NCT07238452
Title: Optimising Pacing Therapy, Integrated Medical Therapy, and Catheter AbLation for Atrial Fibrillation in Heart Failure Trial
Acronym: OPTIMAL AF-HF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jason Andrade, Director, Electrophysiology, Principal Investigator, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-02147
Record Dates: First submitted 2025-05-27; First posted 2025-11-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Atrial Fibrillation (AF)
Keywords: Atrial fibrillation; heart failure; cardiomyopathy; catheter ablation; pulsed field ablation; atrioventricular node ablation; conduction system pacing; cardiac resyncronization therapy
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Optimal Medical Therapy (Active Comparator): Patients randomised to medical rate control will receive evidence-based beta-blockers (extended-release metoprolol succinate, bisoprolol, carvedilol), titrated to achieve a resting heart rate of <100 bpm during AF, in accordance with contemporary guidelines (Appendix B). In the event of patients not achieving satisfactory symptom or heart rate-control with monotherapy, then these agents may be combined with digoxin (trough target 0.5 and 0.9 ng/ml) or oral amiodarone.
  Interventions: Drug: Pharmacological Rate Control
- Catheter Ablation with The Goal of Sinus Rhythm Restoration (Pulmonary Vein Isolation) (Active Comparator): Patients randomised to invasive rhythm control will undergo a percutaneous catheter ablation procedure using standardised techniques to achieve pulmonary vein isolation. The procedure will be performed with a combined radiofrequency + pulsed-field ablation energy catheter. Circumferential lesions around the veins will be considered complete when spontaneous, associated PV potentials are no longer recorded by the circular catheter (entrance block) and when exit block (dissociated spontaneous PV ectopy, and/or local PV capture without conduction from the pulmonary vein into the left atrium) has been demonstrated.
  Interventions: Device: Pulmonary Vein Isolation
- Catheter Ablation with The Goal of Ventricular Rate Control and Regularization (AVJ Ablation) (Active Comparator): Patients randomised to catheter ablation of the AV junction will undergo a percutaneous catheter ablation procedure using standardised techniques to achieve complete AV block. Patients randomised to AVJ ablation will receive a cardiac resynchronisation capable device owing to the risk of pacing induced cardiomyopathy (CRT-D if LVEF ≤35%, CRT-P or CSP with an FDA approved conduction system lead if LVEF 36-40%)
  Interventions: Procedure: Atrioventricular Node Ablation

INTERVENTIONS:
Device: Pulmonary Vein Isolation — PVI
  Arms: Catheter Ablation with The Goal of Sinus Rhythm Restoration (Pulmonary Vein Isolation)
Procedure: Atrioventricular Node Ablation — AVJ
  Arms: Catheter Ablation with The Goal of Ventricular Rate Control and Regularization (AVJ Ablation)
Drug: Pharmacological Rate Control — Rate
  Arms: Optimal Medical Therapy

SUMMARY:
Atrial Fibrillation (AF) and Heart Failure (HF) are colliding global cardiovascular epidemics, individually impairing quality of life and cardiac performance, as well as increasing the risk of hospitalisation and mortality. When AF and HF co-exist, disease progression accelerates and the adverse outcomes are magnified, leading to incrementally higher morbidity, mortality, and healthcare expenditure. The management of AF has been dichotomised into the restoration and maintenance of sinus rhythm ("Rhythm control") or acceptance of AF with control of the ventricular response ("Rate control"). Previous studies suggested that pharmacologic rhythm control and pharmacologic rate control confer similar survival and morbidity outcomes in patients with significant left ventricular dysfunction. Recognising the limitations of pharmacotherapy, more recent studies have examined the utility of catheter ablation procedures, either designed to restore and maintain sinus rhythm (e.g., catheter-based pulmonary vein isolation) or control the ventricular response (e.g., pacemaker implantation in combination with catheter ablation of the atrioventricular junction). Compared to pharmacotherapy, these studies have suggested that catheter ablation may provide sustained improvements in quality of life, decreased hospitalisation and, potentially, improved survival for patients with co-existing AF and HF. However, these studies were performed prior to the modern era of quadruple LV enhancing therapy (beta-blocker, an angiotensin receptor-neprilysin inhibitor, mineralocorticoid receptor antagonist, and an SGLT2 inhibitor). The true impact of catheter-based interventions, and thus the optimal management of AF for patients with co-existing HF is not known. The investigators propose a randomised controlled trial to definitively answer the question regarding the optimal invasive treatment of AF in patients with heart failure with reduced ejection fraction (HFrEF - LVEF ≤ 40%).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older on the date of Informed Consent,
* Atrial fibrillation,
* Left ventricular ejection fraction of 40% or less, measured within 6 months of enrollment,
* Receiving stable foundational HF quadruple therapy at maximally tolerated dose,
* BNP ≥ 100 pg/mL (NT-proBNP ≥ 400 pg/ml), measured within 1 month of randomisation.

Exclusion Criteria:

* Anticipated life expectancy less than one year from the consent date,
* Continuous atrial fibrillation of >1 year in duration,
* Left atrial anteroposterior diameter > 6 cm, volume > 100 mL, or volume index > 60 mL/m2,
* Previous left atrial ablation or left atrial surgery,
* The presence of a percutaneous left atrial appendage closure device,
* Uncontrolled hypo- or hyperthyroidism,
* Subject known to be pregnant or breast-feeding,
* Contraindication to oral anticoagulation therapy,
* Left atrial myxoma,
* Myocardial infarction or percutaneous coronary intervention within 3-months of consent,
* History of, or anticipated to undergo heart transplant, ventricular assist device insertion, or mitral or tricuspid valve repair or replacement within 3-months of the consent date.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2032-12-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular mortality, stroke, and total number of heart failure events | 5 years

SECONDARY OUTCOMES:
Composite of ejection fraction, distance on the 6-minute walk test, and QOL score | 1 year
Time to death from any cause | 5 years
Time to death from cardiovascular cause | 5 years
Number of Participants with unplanned emergency department visit or all-cause hospitalisation | 5 years
Number of Participants with unplanned emergency department visit or hospitalisation for heart failure | 5 years
Number of Participants with unplanned emergency department visit or hospitalisation for atrial fibrillation or arrhythmia | 5 years
Number of Participants with heart failure event | 5 years
Change in Quality of Life from baseline | 5 years
Number of Participants with ischemic stroke or systemic arterial emboli | 5 years
Number of Participants with new onset cognitive dysfunction | 5 years
Change in left ventricular function (ejection fraction) | 5 years
Time to first appropriate and inappropriate ICD intervention (ATP or ICD shock) | 5 years

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD will be decided at a later dat by the academic steering committee.